CLINICAL TRIAL: NCT07085052
Title: Remote Mindfulness Study 2
Brief Title: Remote Mindfulness Training Following Early Life Adversity 2
Acronym: ReMind 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Emily Lindsay, Assistant Professor, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY25020112
Record Dates: First submitted 2025-07-03; First posted 2025-07-25 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Stress; Mindfulness; Early Life Adversity
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness-Based Stress Reduction (MBSR) (Experimental): MBSR is a standardized curriculum-based group program. In this study, MBSR will be adapted to include 10 (rather than the standard 8) weekly 2.5-hour group sessions delivered online, plus a day-long online retreat and 30-45 minutes of home practice assignments six days per week. MBSR includes guided mindfulness meditations intended to foster awareness of present-moment experiences and an open, accepting, and nonjudgmental perspective. Guidance and group discussions also encourage nonjudgmental awareness in everyday life, including when experiencing stress or other challenging emotions. Group discussions involve exploration of habitual reactions to stress and the cultivation of skills such as pausing before responding. Foundationally, the course centers on self-care and group support, including support for the challenge of integrating meditation practice into daily life. Home practice recordings will guide participants through body awareness, mindful movement, and seated meditation.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — 10-week online MBSR program, involving 10 weekly 2.5-hour group sessions, a day-long online retreat, and approximately 45 minutes of home practice assignments six days per week.

SUMMARY:
This pilot study aims to evaluate the effects of a 10-week online Mindfulness-Based Stress Reduction (MBSR) intervention on stress and inflammatory outcomes in a sample of emerging adults with a history of early life adversity. 15 participants (ages 18-29) with a history of childhood trauma will receive online, group-based MBSR sessions over 10 weeks. At pre- and post-intervention, participants will complete laboratory assessments, including self-report questionnaires and blood sample collection to assess markers of inflammation. Data assessing subjective and physiological stress in daily life will be collected for one week at pre- and post-intervention. This preliminary data will be used to test effects of online MBSR on health-relevant outcomes among young adults with a history of childhood trauma.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-29 years
* English speaking
* History of adverse childhood experiences (specifically, moderate-to-severe physical, emotional, or sexual abuse in childhood: scoring >9, >12, or >7 on respective Childhood Trauma Questionnaire subscales)
* Data-enabled Android or iOS smartphone
* Able to meet study requirements

Exclusion Criteria:

* Self-reported diagnosis of chronic physical disease (e.g., cancer, HIV, heart disease, diabetes, bleeding disorder)
* Self-reported diagnosis of chronic mental disorder (e.g., schizophrenia, personality disorder, or psychotic illness), major neurological disorder, or suicidal thoughts or wishes at baseline
* Medication use that interferes with HPA-axis activity (e.g., corticosteroids), autonomic activity (e.g., antihypertensive medication), inflammatory activity (e.g., cholesterol medications), or blood clotting
* Current antibiotic, antiviral, or antimicrobial treatment
* Shift workers
* Pregnancy
* Substance use disorder
* Regular systematic mind-body practice (>2 times per week)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Change in Daily Life Subjective Stress: State Perceived Stress | change in stress assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  State perceived stress assessed in daily life four times per day for one week at two time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Stress will be assessed on a 1-7 Likert scale, with higher scores indicating higher perceived stress.
Change in Daily Life Subjective Stress: Daily Perceived Stress | change in stress assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Daily perceived stress assessed in daily life each evening for one week at two time points via end-of day diary, totaling up to 7 assessments at each time point. All 7 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Stress will be assessed on a 1-7 Likert scale, with higher scores indicating higher perceived stress.
Change in Daily Life Objective Stress: Stress Events in the Past 2.5 Hours | change in stress assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Stress events assessed on a binary scale (yes/no) in daily life four times per day for one week at two time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in logistic MLM analyses. Outcomes will be reported as mean percentage of surveys at each time point that stress events were endorsed, with higher percentages indicating more stress events.
Change in Daily Life Objective Stress: Daily Stress Events | change in stress assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Daily stress events assessed in daily life each evening for one week at two time points via end-of day diary, totaling up to 7 assessments at each time point. All 7 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in logistic MLM analyses. Outcomes will be reported as mean percentage of days at each time point that stress events were endorsed, with higher percentages indicating more stress events.
Change in Daily Life Physiological Stress Reactivity | change in HR reactivity assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Heart Rate (HR) measured continuously in daily life, with HR averaged in 30-minute windows around daily life stress reported via EMA up to four times per day for one week at two time points, totaling up to 28 windows at each time point. All (up to) 28 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Higher scores indicate higher HR in beats per minute (relative to an individual's average daily HR) at high stress moments (relative to an individual's average perceived stress).

SECONDARY OUTCOMES:
Feasibility of Recruitment (Screened Eligible) | assessed pre-enrollment
  Recruitment benchmark: >10% of people screened will be eligible
Feasibility of Recruitment (Enrollment) | assessed at enrollment
  Recruitment benchmark: >60% of those eligible will enroll
Feasibility of Retention | assessed across the entire study period, approximately 14 weeks
  Retention benchmark: >80% retention through intervention and >75% retention through post-intervention assessments
Feasibility of Adherence: MBSR attendance | assessed across the entire 10-week intervention period
  Adherence benchmark: average completion of at least 7 of 11 MBSR sessions
Feasibility of Adherence: Ambulatory Assessments | assessed for 1 week at two time points: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 11 weeks)
  Adherence benchmark: average completion of >75% of ambulatory assessments
Feasibility of Adherence: Mobile Sensor Data | assessed for 1 week at two time points: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 11 weeks)
  Adherence benchmark: collecting Fitbit sensor data on >75% of days
Feasibility of Safe Implementation: Incidence of Treatment-emergent Increases in Mental Health Symptoms | assessed across the entire study period, approximately 14 weeks
  Safety benchmark: <10% of participants showing substantial (>2SD) increases in anxiety, trauma, or depressive symptoms (using PROMIS Anxiety and Depression scales and Posttraumatic Stress Disorder Checklist-Civilian scale described in other outcomes below) combined to create treatment-emergent symptom rate
Acceptability: Treatment Expectancies | assessed in-person at post-intervention laboratory assessment (an average of 13 weeks)
  Acceptability of interventions, with benchmark of >80% of participants giving positive ratings of treatment expectancies (>3 on 6-item Credibility/Expectancy Questionnaire)

OTHER OUTCOMES:
Early Life Adversity: Childhood Trauma | pre-intervention baseline laboratory assessment
  Assessed via the Childhood Trauma Questionnaire (a 28-item scale with three 5-item abuse subscales - physical, sexual, and emotional abuse - ranging from 5-25, with higher scores indicating higher childhood trauma)
Early Life Adversity: Emotional Neglect | pre-intervention baseline laboratory assessment
  Early Life Adversity assessed via the Childhood Experiences of Care and Abuse Inventory (a 16-item scale separated into 8-item mother and father figure emotional neglect subscales ranging from 8-40, with higher scores indicating higher levels of emotional neglect)
Early Life Adversity: Childhood SES Indexed Via Parental Education | pre-intervention baseline laboratory assessment
  Childhood SES indexed via parental educational attainment, ranging from less than high school education to doctoral degree (1 = No High School Diploma, 2 = GED, 3 = High School Diploma, 4 = Technical Training, 5 = Some College, no degree, 6 = Associate Degree, 7 = Bachelor's Degree, 8 = Master's Degree, 9 = MD, PhD, JD, or PharmD), with higher scores indicating higher educational attainment
Early Life Adversity: Childhood SES Indexed by Government Food Assistance | pre-intervention baseline laboratory assessment
  Childhood SES assessed via National Comorbidity Survey: Adolescents item assessing government food assistance
Early Life Adversity: Domestic Violence | pre-intervention baseline laboratory assessment
  Early Life Adversity assessed via Adverse Childhood Experiences Survey (using a 5-item domestic violence subscale, ranging from 0-10, with higher scores indicating higher levels of domestic violence)
Change in Circulating Inflammatory Markers (IL-6) | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Circulating IL-6 assessed via dried blood spot (DBS) [additional funding needed to assess]
Change in Circulating Inflammatory Markers (IL-10) | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Circulating IL-10 assessed via dried blood spot (DBS) [additional funding needed to assess]
Change in Circulating Inflammatory Markers (TNF) | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Circulating TNF assessed via dried blood spot (DBS) [additional funding needed to assess]
Change in Circulating Inflammatory Markers (uPAR) | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Circulating uPAR assessed via dried blood spot (DBS) [additional funding needed to assess]
Change in Circulating Inflammatory Markers (CRP) | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Circulating CRP assessed via dried blood spot (DBS) [additional funding needed to assess]
Change in Daily Life Positive Affect: State | change in affect assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  State positive affect assessed in daily life four times per day for one week at two time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Positive affect will be assessed on a 1-7 Likert scale, with higher scores indicating higher positive affect.
Change in Daily Life Positive Affect: Daily | change in affect assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Daily positive affect (composite of 9 positive affect items across 3 subscales: happiness (happy, pleased, and cheerful), calm (calm, at-ease, and relaxed), and vigor (lively, full-of-pep, and energetic), each assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at two time points via end-of day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Higher scores reflect higher positive affect.
Change in Daily Life Negative Affect: State | change in affect assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  State negative affect assessed in daily life four times per day for one week at two time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Negative affect will be assessed on a 1-7 Likert scale, with higher scores indicating higher negative affect.
Change in Daily Life Negative Affect: Daily | change in affect assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Daily negative affect (composite of 9 negative affect items across 3 subscales: anxiety (on edge, nervous, and tense), depression (sad, depressed, and unhappy), and hostility (hostile, resentful, and angry), each assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at two time points via end-of day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Higher scores reflect higher negative affect.
Change in Daily Life Social Interactions: Interactions in the Past 2.5 Hours | change in interactions assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Number of social interactions assessed in daily life four times per day for one week at two time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Higher numbers indicate more social interactions.
Change in Daily Life Social Interactions: Daily | change in interactions assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Number of social interactions assessed in daily life each evening for one week at two time points via end-of day diary, totaling up to 7 assessments at each time point. All 7 assessments at each of the two time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Higher numbers indicate more social interactions.
Change in Daily Life Mindfulness: Awareness | change in awareness assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Mindful awareness (composite 3-item scale: "Today, I paid attention to what I was doing in the present moment" / "Today, I noticed body sensations come and go" / "Today, I noticed pleasant and unpleasant thoughts and emotions", each item assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at two time points via end- of-day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the two time points (pre- intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Higher composite scores reflect higher mindful awareness.
Change in Daily Life Mindfulness: Acceptance | change in acceptance assessed in daily life for 1 week at two timepoints: pre-intervention ambulatory assessment and post-intervention ambulatory assessment (an average of 11 weeks)
  Mindful acceptance (composite 2-item scale: "Today, I was able to step back and be aware of distressing thoughts, emotions, and sensations, without being taken over by them" / "Today, I did not want to feel the way I was feeling", each item assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at two time points via end- of-day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the two time points (pre- intervention ambulatory assessment, post-intervention ambulatory assessment) will be averaged in MLM analyses. Higher composite scores reflect higher acceptance.
Change in Global Psychosocial Stress: Anxiety | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via PROMIS Anxiety, a 4-item scale with raw scores ranging from 4-20 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t- scores indicating higher anxiety
Change in Global Psychosocial Stress: Depressive Symptoms | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via PROMIS Depression, a 4-item scale with raw scores ranging from 4-20 and converted to t- scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher depressive symptoms
Change in Global Psychosocial Stress: Trauma Symptoms | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via Post-Traumatic Stress Disorder Checklist for Civilians (PCL-C), a 17-item scale ranging from 17-85, with higher scores indicating higher levels of trauma, and scores of 30 or greater indicating at least moderately severe PTSD symptoms
Change in Global Psychosocial Stress: Depersonalization | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via Cambridge Depersonalization Scale (a 29-item scale ranging from 0-116, assessing frequency and duration of depersonalization symptoms, with higher scores indicating greater depersonalization)
Change in Global Psychosocial Stress: Perceived Stress | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via Perceived Stress Scale (a 10-item scale ranging from 0-40, with higher scores indicating higher perceived stress)
Change in Global Psychosocial Stress: Social Isolation | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via PROMIS Social Isolation, a 14-item scale with raw scores ranging from 14 to 70 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher social isolation
Change in Sleep Quality | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via Pittsburgh Sleep Quality Index (6-item short form, ranging from 0-12, with higher scores indicating worse sleep)
Change in Global Psychosocial Resilience: Life Satisfaction | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via PROMIS Life Satisfaction, a 5-item scale with raw scores ranging from 5-35 and converted to t- scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher life satisfaction
Change in Global Psychosocial Resilience: Positive Affect | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via PROMIS Positive Affect, a 15-item scale with raw scores ranging from 15-75 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher positive affect
Change in Global Psychosocial Resilience: Self-Efficacy | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Assessed in-person via PROMIS Self-Efficacy, a 4-item scale with raw scores ranging from 4-20 and converted to t- scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher self-efficacy
Change in Global Mindfulness | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Five Facet Mindfulness Questionnaire-Short Form (a 24-item scale including five subscales - observing, describing, acting with awareness, nonreactivity, and nonjudgment, with average scores ranging from 1-5 and higher scores indicating higher mindfulness)
Change in Global Experiential Avoidance | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Acceptance and Action Questionnaire-II (a 7-item scale ranging from 7-49, with higher scores indicating higher experiential avoidance)
Change in Global Distress Tolerance | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Distress Tolerance Scale (a 15-item scale ranging from 1-5, with higher scores indicating higher distress tolerance)
Change in Global Self-Compassion | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Self-Compassion Scale (a 25-item scale ranging from 1-5, with higher scores indicating higher self-compassion)
Change in Global Interoceptive Awareness | change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 13 weeks)
  Multidimensional Assessment of Interoceptive Awareness Scale (a 32-item scale comprised of eight subscales [Noticing, Not-Distracting, Not-Worrying, Attention Regulation, Emotional Awareness, Self-Regulation, Body Listening, and Trusting] ranging from 0-5, with higher scores indicating greater interoceptive awareness)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Lindsay, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD from this small pilot study.

DOCUMENTS (1):
  • Informed Consent Form (2025-06-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT07085052/ICF_000.pdf